CLINICAL TRIAL: NCT00943124
Title: An Open-Label, Definitive Bioequivalence Study to Compare the Pharmacokinetics of the Simvastatin, Nicotinic Acid, and MK0524 (Laropiprant) Components of a Formulation of MK0524B With That of Zocor™ and MK0524A Tablets
Brief Title: MK0524B Bioequivalence Study (0524B-070)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0524B-070; MK0524B-070; 2009_612
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2010-01-06 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — MK-0524; Simvastatin

ARMS (2):
- MK0524B then Simvastatin + MK0524A (Experimental): Period 1: 1 tablet of MK0524B (ER niacin 900 mg/ laropiprant 20 mg/ simvastatin 20 mg).
  Period 2: 1 tablet of simvastatin 20 mg (Zocor™) and 1 tablet of MK0524A (ER niacin 1000 mg/ laropiprant 20 mg) as separate tablets.
  Interventions: Drug: MK0524B (ER niacin (+) laropiprant (+) simvastatin); Drug: MK0524A (ER niacin + laropiprant); Drug: Simvastatin
- Simvastatin + MK0524A then MK0524B (Experimental): Period 1: 1 tablet of simvastatin 20 mg (Zocor™) and 1 tablet of MK0524A (ER niacin 1000 mg/ laropiprant 20 mg) as separate tablets.
  Period 2: 1 tablet of MK0524B (ER niacin 900 mg/ laropiprant 20 mg/ simvastatin 20 mg).
  Interventions: Drug: MK0524B (ER niacin (+) laropiprant (+) simvastatin); Drug: MK0524A (ER niacin + laropiprant); Drug: Simvastatin

INTERVENTIONS:
Drug: MK0524B (ER niacin (+) laropiprant (+) simvastatin) — Single dose of MK0524B (ER niacin 900 mg/ laropiprant 20 mg/ simvastatin 20 mg) in one of two treatment periods.
  Other Names: MK0524B
Drug: MK0524A (ER niacin + laropiprant) — Single dose of MK0524A (ER niacin 1000 mg/ laropiprant 20 mg) in one of two treatment periods.
  Other Names: MK0524A
Drug: Simvastatin — Single dose simvastatin (Zocor™) 20 mg in one of two treatment periods.
  Other Names: Zocor™

SUMMARY:
This study will evaluate:

1. the bioequivalence of simvastatin and simvastatin acid following dose of simvastatin (ZOCOR™) given together with one tablet of MK0524A or as a component of the triple combination tablet MK0524B.
2. the bioequivalence of laropiprant and ER niacin when administered as the triple combination tablet MK0524B or as the double combination tablet MK0524A given together with simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject is a nonsmoker
* Subject is willing to follow the study guidelines

Exclusion Criteria:

* Subject has or has a history of any illness that might confound the results of the study or make participation in the study unsafe for the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK0524B Then Simvastatin + MK0524A: Period 1: 1 tablet of MK0524B (ER Niacin 900 mg/laropiprant 20 mg/simvastatin 20 mg fixed dose combination tablet).
  Period 2: 1 tablet of simvastatin and 1 tablet of MK0524A (ER Niacin 1000 mg/laropiprant 20 mg) as separate tablets.
- Simvastatin + MK0524A Then MK0524B: Period 1: 1 tablet of simvastatin and 1 tablet of MK0524A (ER Niacin 1000 mg/laropiprant 20 mg) as separate tablets.
  Period 2: 1 tablet of MK0524B (ER Niacin 900 mg/laropiprant 20 mg/simvastatin 20 mg fixed dose combination tablet).
Period: Period 1
Arm/Group | MK0524B Then Simvastatin + MK0524A | Simvastatin + MK0524A Then MK0524B
Started | 110 | 110
Completed | 108 | 108
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Did Not Follow Study Procedures | 1 | 0
Not completed — Personal Reasons | 0 | 1
Period: Period 2
Arm/Group | MK0524B Then Simvastatin + MK0524A | Simvastatin + MK0524A Then MK0524B
Started | 108 | 108
Completed | 108 | 108
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All randomized patients
Arm/Group | Overall Study Population
Number analyzed (Participants) | 220
Age, Continuous [Mean (Full Range); unit: years] | 35.11 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 128
Height [Mean (Full Range); unit: Centimeters] | 169.58 [147 to 193]
Weight [Mean (Full Range); unit: Kilograms] | 72.99 [43.6 to 111.2]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Area Under the Curve (AUC(0 to 48hr)) for Simvastatin Acid
Description: Plasma Area Under the Curve of simvastatin acid, the active metabolite of simvastatin
Time Frame: Through 48 Hours Post Dose
Population: Two hundred-twenty (220) subjects were enrolled in this study. Due to early dropout (N=4), mis-handling of plasma samples (N=10) and the limitation of the assay (N=10), data from a total of 200 and 202 subjects were available for simvastatin acid AUC(0 to 48 hour) analysis for MK0524B and Simvastatin + MK0524A, respectively.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL * Hour
Groups:
- MK0524B: MK0524B: 1 tablet of ER Niacin 900 mg/laropiprant 20 mg/simvastatin 20 mg fixed dose combination tablet.
- Simvastatin + MK0524A: Simvastatin + MK0524A : 1 tablet of simvastatin 20 mg (ZOCOR) and 1 tablet of MK0524A (ER Niacin 1000 mg/laropiprant 20 mg) as separate tablets
Arm/Group | MK0524B | Simvastatin + MK0524A
Number analyzed (Participants) | 200 | 202
ng/mL * Hour | 9.19 (8.38) | 8.03 (7.78)
Statistical Analysis 1: Comparison: MK0524B vs Simvastatin + MK0524A; Least-Squares Mean Ratio (Fixed Dose Combination (FDC)/Co-administration); Test type: Non-Inferiority or Equivalence — Power: If the true geometric mean ratio (GMR MK0524B/Simvastatin + MK0524A) is 1.00 for all the eight primary endpoints, then a sample size of N=220 subjects provides this study with greater than 99.2% probability of observing the 90% confidence intervals (CIs) of all the eight endpoints to be contained within [0.80, 1.25], assuming nonnegative associations among the 8 endpoints; Least-Squares Mean Ratio = 1.14, 90% CI [1.09 to 1.20]

2. Primary Outcome: Peak Plasma Concentration (Cmax) of Simvastatin Acid
Description: Peak Plasma Concentration (Cmax) for Simvastatin Acid, the active metabolite of simvastatin
Time Frame: 48 Hours Post Dose
Population: Two hundred-twenty (220) subjects were enrolled in this study. Due to early dropout (N=4), mis-handling of plasma samples (N=10) and the limitation of the assay (N=10), data from a total of 201 and 202 subjects were available for simvastatin acid Cmax analysis for MK0524B and Simvastatin + MK0524A, respectively.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | MK0524B | Simvastatin + MK0524A
Number analyzed (Participants) | 201 | 202
ng/mL | 1.016 (0.946) | 0.918 (0.906)
Statistical Analysis 1: Comparison: MK0524B vs Simvastatin + MK0524A; Least-Squares Mean Ratio (Fixed Dose Combination (FDC)/Co-administration); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least-Squares Mean Ratio = 1.11, 90% CI [1.05 to 1.16]

3. Primary Outcome: Plasma Area Under the Curve (AUC(0 to 48 Hour)) for Simvastatin
Description: Plasma Area Under the Curve of simvastatin
Time Frame: Through 48 Hours Post Dose
Population: Two hundred-twenty (220) subjects were enrolled in this study. Due to early dropout (N=4), mis-handling of plasma samples (N=2) and the limitation of the assay (N=10), data from a total of 208 and 210 subjects were available for simvastatin AUC(0-48 hour) analysis for MK0524B and Simvastatin + MK0524A, respectively.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL * Hour
Arm/Group | MK0524B | Simvastatin + MK0524A
Number analyzed (Participants) | 208 | 210
ng/mL * Hour | 15.03 (9.88) | 15.56 (9.11)
Statistical Analysis 1: Comparison: MK0524B vs Simvastatin + MK0524A; Least-Squares Mean Ratio (Fixed Dose Combination (FDC)/Co-administration); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least-Squares Mean Ratio = 0.97, 90% CI [0.93 to 1.00]

4. Primary Outcome: Peak Plasma Concentration (Cmax) of Simvastatin
Time Frame: 48 Hours Post Dose
Population: Two hundred-twenty (220) subjects were enrolled in this study. Due to early dropout (N=4), mis-handling of plasma samples (N=2) and the limitation of the assay (N=10), data from a total of 209 and 210 subjects were available for simvastatin Cmax analysis for MK0524B and Simvastatin + MK0524A, respectively.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | MK0524B | Simvastatin + MK0524A
Number analyzed (Participants) | 209 | 210
ng/mL | 5.81 (4.31) | 6.33 (4.64)
Statistical Analysis 1: Comparison: MK0524B vs Simvastatin + MK0524A; Least-Squares Mean Ratio (Fixed Dose Combination (FDC)/Co-administration); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least-Squares Mean Ratio = 0.92, 90% CI [0.87 to 0.97]

5. Primary Outcome: Plasma Area Under the Curve (AUC(0 to Infinity)) for Laropiprant
Description: Plasma Area Under the Curve of Laropiprant
Time Frame: 48 Hours Post Dose
Population: Two hundred-twenty (220) subjects were enrolled in this study. Due to early dropout (N=4), data from a total of 217 and 216 subjects were available for laropiprant AUC(0 to infinity) analysis for MK0524B and Simvastatin + MK0524A, respectively
Measure: Least Squares Mean (Standard Deviation); unit: nmol/L * hour
Arm/Group | MK0524B | Simvastatin + MK0524A
Number analyzed (Participants) | 217 | 216
nmol/L * hour | 5486 (2832) | 5405 (2618)
Statistical Analysis 1: Comparison: MK0524B vs Simvastatin + MK0524A; Least-Squares Mean Ratio (Fixed Dose Combination (FDC)/Co-administration); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least-Squares Mean Ratio = 1.02, 90% CI [0.99 to 1.04]

6. Primary Outcome: Peak Plasma Concentration (Cmax) of Laropiprant
Time Frame: 48 Hours Post Dose
Population: Two hundred-twenty (220) subjects were enrolled in this study. Due to early dropout (N=4), data from a total of 217 and 216 subjects were available for laropiprant Cmax analysis for MK0524B and Simvastatin + MK0524A, respectively
Measure: Least Squares Mean (Standard Deviation); unit: nmol/L
Arm/Group | MK0524B | Simvastatin + MK0524A
Number analyzed (Participants) | 217 | 216
nmol/L | 1030 (642) | 953 (542)
Statistical Analysis 1: Comparison: MK0524B vs Simvastatin + MK0524A; Least-Squares Mean Ratio (Fixed Dose Combination (FDC)/Co-administration); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least-Squares Mean Ratio = 1.08, 90% CI [1.02 to 1.14]

7. Primary Outcome: Peak Plasma Concentration (Cmax) of Nicotinuric Acid
Description: Peak Plasma Concentration (Cmax) for Nicotinuric Acid, one of the active metabolites of Niacin
Time Frame: 24 Hours Post Dose
Population: Two hundred-twenty (220) subjects were enrolled in this study. Due to early dropout (N=4) and missing samples (N=1), data from a total of 215 and 216 subjects available for plasma nicotinuric acid analysis for MK0524B and Simvastatin + MK0524A, respectively.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | MK0524B | Simvastatin + MK0524A
Number analyzed (Participants) | 215 | 216
ng/mL | 620 (536) | 807 (469)
Statistical Analysis 1: Comparison: MK0524B vs Simvastatin + MK0524A; Least-Squares Mean Ratio (Fixed Dose Combination (FDC)/Co-administration); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least-Squares Mean Ratio = 0.77, 90% CI [0.72 to 0.82]

8. Primary Outcome: Total Urinary Excretion of Niacin and Its Metabolites
Time Frame: 96 Hours Post Dose
Population: Two hundred-twenty (220) subjects were enrolled in this study. Due to early dropout (N=4), data from a total of 216 subjects were available for both MK0524B and Simvastatin + MK0524A for analysis of urinary excretion of nicotinuric acid and metabolites
Measure: Least Squares Mean (Standard Deviation); unit: µmol
Arm/Group | MK0524B | Simvastatin + MK0524A
Number analyzed (Participants) | 216 | 216
µmol | 5339 (968) | 5825 (1188)
Statistical Analysis 1: Comparison: MK0524B vs Simvastatin + MK0524A; Least-Squares Mean Ratio (Fixed Dose Combination (FDC)/Co-administration); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least-Squares Mean Ratio = 0.92, 90% CI [0.89 to 0.94]

ADVERSE EVENTS:
Description: Although a subject/patient may have had two or more clinical adverse experiences, the subject/patient is counted only once within a category. The same subject/patient may appear in different categories.
Arm/Group | MK0524B | Simvastatin + MK0524A
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/220
Other Adverse Events (participants affected / at risk) | 61/220 | 58/220
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK0524B (N=220) | Simvastatin + MK0524A (N=220)
Palpitations (Cardiac disorders) | 0 | 1
Ear Discomfort (Ear and labyrinth disorders) | 1 | 3
Ocular Hyperaemia (Eye disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 7 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 0
Chapped Lips (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Eructation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 15 | 12
Salivary Hypersecretion (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 5
Fatigue (General disorders) | 1 | 0
Feeling Hot (General disorders) | 3 | 2
Feeling Jittery (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Burning Sensation (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 9 | 17
Migraine (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 4 | 3
Somnolence (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Syncope Vasovagal (Nervous system disorders) | 1 | 2
Hypervigilance (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 3
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 8 | 17
Vasodilatation (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.